CLINICAL TRIAL: NCT06069011
Title: Improving Access to Quality Care for Children and Adolescents Presenting to the Pediatric Emergency Department With Musculoskeletal Problems: a Pilot Randomized Control Trial
Brief Title: Direct Access Physiotherapy in the Pediatric Emergency Department
Acronym: PedEDmsk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Senior Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-9673
Record Dates: First submitted 2023-09-11; First posted 2023-10-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Pain; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary (Experimental): Interdisciplinary model for management of low acuity msk complaint
  Interventions: Other: Interdisciplinary management
- Usual care (Active Comparator): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Other: Interdisciplinary management — assessment and treatment in an interdisciplinary model
  Arms: Interdisciplinary
Other: usual care — assessment and treatment in usual care model
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to compare two methods of managing low acuity musculoskeletal complaints in children and adolescents ages 6 to 17.99 years in the pediatric emergency department. The main question it aims to answer is whether delivering care in two methods is feasible. Participants will receive care while in the emergency department and will be followed for a period of 1-month post-presentation.

ELIGIBILITY:
Inclusion Criteria:

* aged 6.00-17.99 years of age
* present to the Montreal Children's Hospital Emergency Department with a suspected MSK complaint, traumatic or not
* are given a triage score of 3 (urgent), 4 (less urgent), or 5 (nonurgent) according to the Canadian Triage and Acuity Scale (CTAS)
* are able to communicate in French or English

Exclusion Criteria:

* present with a major MSK condition requiring urgent care (e.g., open fracture, open wound)
* a red flag (e.g. progressive neurological disorder, infectious symptoms)
* a co-morbid unstable condition.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of consent | through study completion an average of 4 weeks post-enrolment
  rate of consented patients related to patients approached rate of randomization, feasibility of administration of outcomes
Completed outcome measures | through study completion an average of 4 weeks post-enrolment
  proportion of participants who complete all outcome measures

SECONDARY OUTCOMES:
Pain intensity on faces rating scale | through study completion an average of 4 weeks post-enrolment
  Pain intensity on faces rating scale, scale from 0 to 10, with 10 being a worse score
Pain interference with function PROMIS scale | through study completion an average of 4 weeks post-enrolment
  PROMIS Pediatric Pain Interference - Short Form 8a, 8 items scores from 1-5 with 5 being a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No